CLINICAL TRIAL: NCT05935670
Title: Passive Limb Movement Study
Acronym: PLM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Matthew J. Durand, Associate Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PRO00047520
Record Dates: First submitted 2023-06-22; First posted 2023-07-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Stroke; Vascular Diseases; Ischemic
Keywords: Ischemic Conditioning; Blood Flow; Peripheral Microvascular Function; Neuromuscular Function
MeSH Terms: conditions — Stroke; Vascular Diseases; Ischemia

STUDY DESIGN:
Intervention Model Description: The investigators will enroll and complete visits for 55 individuals within the study including individuals post-stroke (n = 20), their age- and sex-matched controls (CON, n = 20), and young healthy controls (CONyoung, n = 15). This study includes 2 visits to the Athletic and Human Performance Research Center (AHPRC) at Marquette University. The investigators will measure femoral blood flow to passive limb movement and active contractions pre-/post- ischemic conditioning high (225 mmHg) and ischemic conditioning low (25 mmHg).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Ischemic Conditioning - High (Experimental): During each testing session, the investigators will be measuring how one treatment of ischemic conditioning effects leg blood flow and muscle function. One day participants will receive a high cuff inflation pressure on the leg, called ischemic conditioning - high (225 mmHg).
  Interventions: Device: Ischemic Conditioning
- Ischemic Conditioning - Low (Experimental): During each testing session, the investigators will be measuring how one treatment of ischemic conditioning effects leg blood flow and muscle function. One day participants will receive a low cuff inflation pressure on the leg, called ischemic conditioning - low (25 mmHg).
  Interventions: Device: Ischemic Conditioning

INTERVENTIONS:
Device: Ischemic Conditioning — The cuff will be placed around the proximal, paretic thigh (or dominant thigh for controls) and inflated for 5 minutes in a supine or semi-reclined position, then released for a 5-minute recovery period. Five cycles of inflation and recovery will be performed (45 minutes total).These inflations will be done using a cuff similar to what is used for taking blood pressure.

SUMMARY:
Stroke survivors have compromised vascular function which may contribute to secondary stroke risk, cardiovascular disease, and may limit their exercise tolerance. No studies have examined how femoral blood flow responds to both passive leg movement, a measure of microvascular function, as well as active leg contractions, a measure of the hyperemic response to exercise. Leg muscles with a reduced blood flow response to movement could be associated with decreased neuromuscular function, such as leg strength and fatigue. Preliminary data showing a single bout of ischemic conditioning may improve vascular function and muscle activation in healthy adults and individuals post-stroke. Therefore, the investigators want to examine if ischemic conditioning will also improve the blood flow response to passive leg movements as well as during single leg active contractions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals Post-Stroke

  * 18 - 85 years of age
  * Cortical or sub-cortical stroke ≥ 6 months ago with residual hemiparesis
  * Able to give informed consent and follow 2-step command.
  * English Speaking
* Age- and Sex-Matched Controls (CON)

  * Matched to age of individual post- stroke ± 5 years.
  * Matched to sex of individual post-stroke
  * Able to give informed consent and follow 2-step command.
  * English Speaking
* Young Healthy Adults (CONyoung)

  * Age 18-30 years old
  * Able to give informed consent and follow 2-step command.
  * English Speaking

Exclusion Criteria:

* All Groups

  * Unable to stand from chair and walk 10 meters without physical assistance from another person (able to use assistive device).
  * History of blood clots in the extremities or any condition in which compression of the thigh or transient ischemia is contraindicated (i.e., wounds in the leg).
  * Chronic lasting symptoms (> 6 months) of severe COVID-19 (i.e., hospitalization)
  * Low back or hip pain that limits lower extremity motor testing.
  * History of head trauma or concussion within the past 6 months
  * Comorbid neurological disorder
  * Peripheral vascular disease
  * Myocardial infarction in the previous year
  * Condition where fatiguing contractions or resisted leg contractions are contraindicated
  * Resting SBP ≥180 mmHg or DBP ≥ 100 mmHg
  * Pregnancy or breastfeeding.
  * Other significant medical condition likely to influence study or jeopardize safety as assessed by the Primary Investigator
* CON and CONyoung

  * History of Stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ultrasound Measured Femoral Blood Flow during Passive Limb Movement (PLM) | Change from Baseline PLM Femoral Blood Flow after IC (3 hours)
  Microvascular response to single passive leg movement
Ultrasound Measured Femoral Blood Flow during Active Limb Contraction | Change from Baseline MVCs Femoral Blood Flow after IC (3 hours)
  Hyperemic Response to Maximal Voluntary Contractions (MVCs)

SECONDARY OUTCOMES:
Ultrasound measured Femoral Blood Flow following Neuromuscular Fatigue Task | Post Ischemic Conditioning (15 minutes)
  Hyperemic Response to Fatiguing Muscle Contractions

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Durand, PhD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No